CLINICAL TRIAL: NCT05416216
Title: Wellbeing of the ECE Workforce in Low-resourced Locations
Acronym: WELL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado School of Public Health (Other)
Responsible Party: Principal Investigator, Charlotte Farewell, Assistant Professor, Colorado School of Public Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 21-4662
Record Dates: First submitted 2022-06-06; First posted 2022-06-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Burnout, Caregiver; Stress; Mental Health Wellness
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomized Trial. To evaluate the effectiveness of the WELL intervention the researchers will implement a stepped wedge cluster randomized trial. In this design, ECE centers (steps 1-3) start the trial at the same point in time and act as controls until they are randomized to crossover from control to intervention conditions. This design has been used for pragmatic public health trials conducted as part of routine practice where phased implementation is preferable for feasibility and when the interventions are expected to provide more good than harm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In the stepped wedge design, ECE centers start the trial at the same point in time and act as controls with no intervention until they are randomized to crossover from control to intervention conditions.
- WELL intervention (Experimental): 'WELL intervention' is when implementation of the one-year, three-strategy WELL intervention begins (see description).
  Interventions: Behavioral: WELL

INTERVENTIONS:
Behavioral: WELL — The WELL intervention is a multi-level, three-strategy program to promote the wellbeing of the ECE workforce.
  Arms: WELL intervention

SUMMARY:
The WELL program is a multi-strategy early childhood education (ECE) center-based intervention focused on ensuring that formal ECE providers prioritize their own self-care and well-being and have access to resources and supports that improve their skills to have stable and responsive relationships with young children in their care.

The overarching goals of this proposed project include:

* To utilize Head Start-University partnerships to investigate constructs within the National Institute of Occupational Safety and Health (NIOSH) Worker Wellbeing framework (e.g., Workplace Physical Environment and Safety Climate, Workplace Policies and Culture) among Head Start staff (n=360 Head Start staff) that are most associated with overall well-being.
* To adapt and refine the WELL program to target specific constructs that are most significantly related to overall well-being among the ECE workforce identified in Aim 1 and then to test the effectiveness of WELL (n=36 Head Start centers; n=360 Head Start staff).
* To collect data to inform the implementation and dissemination of the WELL project research findings and products and initiate translation activities to achieve large-scale adoption.

DETAILED DESCRIPTION:
To evaluate the effectiveness of the WELL intervention on our primary outcome (well-being) and secondary outcomes (turnover, burnout, quality of caregiver-child relationship, and child social-emotional development), the researchers will implement a stepped wedge cluster randomized trial with 3 cohorts including approximately 12 ECE centers/cohort (Head Start classrooms with birth - 5-year-olds) (10 Head Start staff/center). In the stepped wedge design, ECE centers (steps 1-3) start the trial at the same point in time and act as controls until they are randomized to crossover from control to intervention conditions. This design has been used for pragmatic public health trials conducted as part of routine practice where phased implementation is preferable for feasibility and when the interventions are expected to provide more good than harm. In the context of community-based participatory research, it allows all participating communities to receive the intervention. It also maximizes statistical power compared with a parallel cluster randomized design because the intervention effect is estimated not only between cluster comparisons but also within cluster comparisons. There are five phases for the study. 1) 'Control' is when the ECE centers receive standard health promotion/professional development opportunities. The team will document 'usual care' during the control periods. 2) 'WELL intervention' is when implementation of the three-strategy WELL intervention begins. 3) 'Plan for sustainability' is the year allocated to plan for how the project infrastructures and activities will be sustained once research support/funding is completed. Follow-up technical assistance will be offered in this year, but it will be much less intensive than during the intervention implementation year. 4) 'Sustaining WELL' is the first phase of withdrawal of research intervention support, drawing on plans for supplemental funding identified, while maintaining support for research data collection. 5) 'Observing sustainability at a distance' is the last phase and involves withdrawal of all funding supports for ECEs and operating expenses while observing the implementation and sustainability of WELL intervention.

WELL INTERVENTION

The 3-strategy intervention includes:

Strategy 1. Organization-Level: WELL PSE Change Process. Implementing policy, system and environment (PSE) changes in ECE settings can play a key role in promoting ECE provider well-being because these are more likely to be sustained over time.51 The WELL PSE Change Process is a strategic planning process that is an adaptation of Intervention Mapping and is aligned with community-based participatory research principles.27 The PSE Change Process involves convening an ECE center-specific interdisciplinary team comprised of an average of five members including ECE teachers, directors, education supervisors, and human resources staff. A WELL Program Interventionist will lead the team through one-hour meetings on a monthly basis (5-7 meetings) and utilize three change-making strategies to implement PSE changes in the ECE setting: 1) conduct a strengths and needs assessment of their center using a menu of evidence-based PSE changes related to a specific outcome (e.g. worker well-being), 2) prioritize potential PSE changes based on importance and feasibility, and 3) develop action plans with specific action steps for implementation and sustainability of their highest priority PSE changes. The menu of best practices will include PSE changes associated with the domains of the Worker Well-being Framework that were identified as being most significantly related to overall well-being in Aim 1. Examples of PSE change options and alignment with specific worker well-being domains include relaxation breaks built into the daily schedule (Health Status), updated organizational policy highlighting commitment to health and safety (Workplace Policies and Culture), and leadership trainings for supervisors (Work Evaluation and Experience) (n=4 PSE changes/center).

Strategy 2. Interpersonal-Level: WELL Social Support Activities. Social support is consistently linked to good mental health, in part because supportive actions buffer stress. The WELL intervention will include several group-based health-promotion activities that increase social support and networking opportunities among Head Start teachers and between Head Start teachers and management. These workplace well-being group activities will be implemented twice/year and will directly link to the PSE changes selected by Head Start settings. They will aim to increase leadership support and communication, teamwork and respect in the workplace, which have been shown to be related to ECE workforce well-being. Examples of social networking activities include: group-based walking and mindfulness challenges to foster workplace health climate. Additionally, a center-specific Wellness Champion (WC) will be identified to support coordination of these activities and encourage staff buy-in and engagement and give out incentives for participation (e.g., yoga mats, water bottles). A person-centered social network analysis will be conducted with ECE caregivers in each center to understand the internal social network of a center and to inform the social connection activities.

Strategy 3. Individual-Level Supports: Self-Care Plan, mWELL and Lunch and Learn Sessions: Before the implementation of the WELL PSE Change Process, the ECE staff will participate in a facilitated group training (at pre-service) that will introduce the concept of self-care and will walk each ECE provider through the creation of their individualized self-care plan with SMART goals. The self-care plan will cover the following areas: relationship to self; relationship to others; relationship to environment; relationship to caregiver role; and relationship to technology. Following the completion of their self-care plan, the ECE providers will be invited to enroll in the mobile WELL (mWELL) program, a free text messaging program that will promote self-care and mindfulness practices. Mobile health (mHealth)-based interventions delivered through text messaging are becoming more widely used to promote well-being. The mWELL program will be based on the Theory of Planned Behavior (TPB), a theory that focuses on behavioral intent based on an individual's perceived ability to exert self-control. There will be 4 text message cycles for a single program year. Each message cycle will contain 30 core text messages that address the following themes (in this order): self-care, mindfulness practices, well-being related to the caregiving role, and activities for promoting high-quality relationships with children. Each theme will contain approximately 7-8 text messages and 2-3 study text messages. Theme texts will be aligned with the mWELL logic model and based on the theoretical constructs of knowledge, attitudes, subjective norms, perceived behavioral control, intention, and behavior. Participants will receive an average of two text messages every week. The messages will be simple and include goal setting for self-care changes, mindfulness activities, tips specific to caregiver well-being promotion, and links to Head Start staff-specific resources.

The last WELL program strategy to promote individual-level behavior change related to self-care and well-being promotion will be the Lunch and Learn (L&L) sessions (n=4/center) and monthly newsletters for all Head Start staff that focus on each of the PSE changes and associated worker well-being domains identified by the wellness teams, including, and not limited to: workplace design, discrimination, work stress, mental health, and organizational support for work/life balance. The sessions will be based on what is learned in Aim 1 and will consist of 30-minute workshops comprised of both didactic and experiential activities led by the WELL Program Interventionist and will support full implementation and dissemination of the well-being-related changes throughout the ECE setting.

ELIGIBILITY:
Inclusion Criteria:

* Early childcare education providers employed in one of five Head Start-funded ECE centers in Colorado who are providing care for children ages 0-5
* Aged 18 years or older

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Early care and Education Worker Wellbeing | Pre-Post Years 1-5
  Measured as a latent construct via a 68-item National Institute of Occupational Safety and Health Worker Wellbeing Questionnaire that encompasses 5 domains (work evaluation and experience, work safety and physical climate, work policies and culture, health status, and home community and society). The scale total ranges from 0-68 with higher scores indicating higher well-being

SECONDARY OUTCOMES:
Burnout | Pre-Post Years 1-5
  Measured quantitatively via the 22-item Maslach Burnout Inventory Survey. The scale ranges from 0 to 132 with higher scores indicating higher levels of burnout.
Turnover Intent | Pre-Post Years 1-5
  Measured quantitatively via 2-items from the Turnover Intent Scale. Scores range from 2 to 10 with higher scores indicating higher turnover intent.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Adams County Head Start, Brighton, Colorado
  - Denver Great Kids Head Start, Denver, Colorado
  - Otero Junior College Head Start, La Junta, Colorado
  - Jefferson County Head Start, Lakewood, Colorado
  - Lakewood Head Start, Lakewood, Colorado

IPD SHARING:
Plan to Share IPD: No